CLINICAL TRIAL: NCT06276465
Title: Combination of Darolutamide and Stereotactic Body Radiation Therapy in Patients With Castration Resistant Prostate Cancer and Oligometastases on Functional Imaging
Brief Title: Treatment With Darolutamide +/- Radiation Therapy for Patients With a Castration Resistant Cancer and Metastases Detected by Functional Imaging
Acronym: PEACE8
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GTG-2306; 2023-507482-26-00 (Other: EU-CT)
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Prostatic Cancer, Castration-Resistant
Keywords: Phase 3; International; Multicentric; Randomised; Stereotactic body radiation therapy (SBRT); PET-PSMA; mCRPC; nmCRPC; CRPC; oligometastases; functional imaging; darolutamide
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — darolutamide; Radiosurgery; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly allocated in a 1:1 ratio to either the:
  * Control arm: ADT + darolutamide.
  * Experimental arm: ADT + darolutamide + SBRT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT + darolutamide (Active Comparator): Up to 5 years of treatment
  Interventions: Drug: Darolutamide 300 mg; Drug: Androgen deprivation therapy
- ADT + darolutamide + SBRT (Experimental): Up to 5 years of treatment
  Interventions: Drug: Darolutamide 300 mg; Radiation: Stereotactic body radiation therapy; Drug: Androgen deprivation therapy

INTERVENTIONS:
Drug: Darolutamide 300 mg — 2 tablets of 300 mg twice daily (=1200 mg/day) up to 5 years from randomisation
  Other Names: Nubeqa
Radiation: Stereotactic body radiation therapy — Over one week,30 Gy in 3 fractions of 10 Gy
  Other Names: SBRT
  Arms: ADT + darolutamide + SBRT
Drug: Androgen deprivation therapy — Continuous ADT during the study course. The choice of ADT is left to the discretion of the investigator.
  Other Names: ADT

SUMMARY:
In earlier stages of prostate cancer, male sexual hormones (androgens) stimulate the growth of cancer cells. Castration-resistant prostate cancer (CRPC) means that the prostate cancer continued to grow despite patients are taking hormone therapy to control the disease. One of the standard treatments for these patients is so-called 'new generation' hormonal therapy. These hormone therapies include apalutamide, enzalutamide, or darolutamide. They work by blocking androgen receptors that play an important role in the growth of prostate cancer.

In the case of oligometastatic CRPC, the cancer has gone beyond the prostate and has spread to other organs in the body (metastases), but these metastases remain limited in number.

An early detection of the oligometastatic CRPC and appropriate treatment may prolong survival in these patients.

The treatment proposed as part of this research is a combination of oral darolutamide, approved in Europe to treat patients with CRPC who do not have metastasis visible on CT-scan or bone scintigraphy (but visible with positron emission tomography-scan (PET-Scan), a more precise imaging technique) with stereotactic body radiotherapy (SBRT), a new radiotherapy technique guided by very high precision medical imaging. This method makes it possible to better target cancer cells while preserving neighboring healthy organs.

The principal objective of this trial is to evaluate the efficacy of the combination of SBRT with darolutamide, compared to darolutamide.

DETAILED DESCRIPTION:
PEACE 8 is a phase III open-label, randomised (patients are randomly assigned to treatment), international, multicentre trial, evaluating the benefit of adding SBRT to darolutamide for treating patients with oligometastatic CRPC.

Eligible patients will be randomised into either an experimental group receiving darolutamide + SBRT or a control group receiving darolutamide. In both arms, all patients will receive continuous castration (ADT) during the trial course.

Patients' participation in the trial will not exceed 60 months after randomisation, including a maximum treatment duration of 60 months and follow-up up to 60 months after randomisation.

After signing the consent form, patients will enter the pre-inclusion period (before the start of treatment), during which the investigator will carried out all the tests required to assess their eligibility, including demographic data collection, tumour evaluation, and clinical and biological assessments.

Patients will receive doralutamide until disease progression or unacceptable toxicity for a maximum of 5 years after the start of treatment.

To receive treatment, the patient will need to go to hospital, where, at each visit, the medical team will conduct medical examinations before administering the treatment to assess the patient's general state of health and tolerance to the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Patients aged ≥18 years.
3. Patient with histologically confirmed of adenocarcinoma prostate cancer without small cell or pure endocrine features.
4. Patient with a history of local treatment with curative intent for localised prostate cancer, including surgery or radiotherapy.
5. Patients with castration resistant prostate cancer, defined as either:

   * An increasing PSA level, confirmed in 3 consecutive assessments performed at least 1 week apart. This despite androgen deprivation therapy and castrate levels of testosterone.
   * Tumour progression of soft tissue according to the response criteria in solid tumours (RECIST) version (v)1.1.
   * Tumour progression on bone scan, according to PCWG3 criteria.

   N.B. The two latter conditions only apply to the M1CRPC population.
6. Detection of 1 to 5 metastatic sites (pelvic lymph nodes included) on new generation PET using either choline, fluciclovine, or PSMA as tracer.
7. All metastatic sites must be amenable to stereotactic radiation therapy.
8. Patient with normal haematological function: absolute neutrophil count (ANC) >1.0 x 10⁹/L, platelets count ≥100 x 10⁹/L, and haemoglobin ≥9.0 g/dL.
9. Patient with normal liver function with total bilirubin ≤1.5 upper limit of normal (ULN) (unless documented Gilbert's syndrome), aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤2.5 ULN (≤5 ULN in the presence of liver metastases).
10. Adequate liver function with bilirubin <3 mg/dL and albumin >2.5 g/dL.
11. Systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg, as documented at baseline. Patients with hypertension are eligible if their hypertension is controlled and they meet all other eligibility criteria.
12. Adequate kidney function with a creatinine clearance >30 mL/min (Cockcroft-Gault).
13. Patient with Eastern Cooperative Oncology group (ECOG) performance status (PS) ≤1.
14. Patient is willing to use contraceptive during and for at least 1 week after discontinuing darolutamide.
15. Patient affiliated to the social security system (or equivalent according to local regulations for participation in clinical trials).
16. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

1. Patient previously treated for metastatic prostate cancer with a novel hormonal agent (NHA), a CYP17 inhibitor, ketoconazole, chemotherapy, or immunotherapy.
2. A history of cancer, other than the prostate cancer under study, within the 3 years prior to study inclusion, excluding cured localised cancer such as non-melanomatous skin cancer and non-muscle invasive bladder cancer.
3. Presence of an uncontrolled disease or affection that according to the investigator will hinder compliance with the trial procedures or requires hospitalisation.
4. Known to have active viral hepatitis, active human immunodeficiency virus (HIV) A at screening.
5. Patients with known allergy or severe hypersensitivity to the study treatment or any of its excipients.
6. Inability to swallow oral medications.
7. Gastrointestinal disorder or procedure that can be expected to interfere significantly with the absorption of study treatment.
8. Any of the following within 6 months before randomisation: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft; congestive heart failure New York Heart Association (NYHA) Class III or IV.
9. Patients participating in another therapeutic trial within the 30 days prior to randomisation.
10. Patients unable to comply with trial obligations for geographic, social, or physical reasons, or who are unable to understand the purpose and procedures of the trial.
11. Person deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2029-10-15 (Estimated); Study Completion 2032-10-07 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-free survival (rPFS) | From randomization to disease progression or death, up to 5 years.
  The radiographic Progression-free survival is defined as the time interval between the randomisation and radiographic disease progression with conventional imaging (CT-scan or bone-scan), or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Time to treatment failure (TTF) | From randomization to discontinuation of darolutamide, up to 5 years
  The time to treatment failure is defined as the time interval between randomisation and the discontinuation of darolutamide, irrespective of the reason for discontinuation.
Overall survival (OS) | From randomization to death from any cause, up to 5 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Prostate cancer-specific survival | From randomization to death due to prostate cancer, up to 5 years.
  The prostate cancer-specific survival is defined as the time interval between randomisation and the date of death due to prostate cancer.
Time to PSA progression | From randomization to PSA progression, up to 5 years.
  The time to PSA progression is defined as the time interval between the date of randomisation and the date of PSA progression. PSA progression is defined, in accordance with the PCWG3 guidelines which retained the PCWG2 definition (2007 guidelines).
Biochemical response rate | Throughout study completion, up to 5 years.
  The biochemical response rate is defined as the proportion of patients with a decrease in PSA levels of ≥50% from baseline levels.
Time to next symptomatic skeletal event (SSE) | Time from randomization to the first symptomatic skeletal event, up to 5 years.
  The time to next symptomatic skeletal event is defined as the time interval from randomisation until the first occurrence of a symptomatic fracture, bone radiation (for pain or neurological complication), bone surgery (for pain or neurological complication), or spinal cord compression.
Time to pain progression | Time from randomization to the first occurence of pain progression, up to 5 years.
  The time to pain progression is defined as the time interval from randomisation until the first occurrence of any of the following:
  * Increase of ≥2 points, from baseline, in question 3 of the Brief Pain Inventory-Short Form (BPI-SF) questionnaire (item related to the worst pain in the last 24 hours).
  * Initiation of opioid treatment for cancer pain.
  * Increase in the use of opioid treatment of ≥30% in terms of frequency of use or cumulative dose.
Safety/tolerance | Throughout study completion, up to 5 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Functional Assessment of CAncer Therapy - Prostate (FACT-P) | At baseline, 1 month, every 4 months during treatment period, and at the end of treatment (up to 5 years).
  The FACT-P is a self-assessment questionnaire to estimate the health-related quality of life in men with prostate cancer. This questionnaire, composed of 39 items consists of four subscales: Physical Well-Being (7 items), Social/Family Well-Being (7 items), Emotional Well-Being (6 items), Functional Well-Being (7 items), and prostate cancer subscale (12 items). Subscales are rated on 5-point Likert-type scale (from 0 = "Not at all" to 4 = "Very much"). For all subscales, a higher score represents better quality of life.
Brief Pain Inventory - Short Form (BP-SFI) questionnaire | At baseline, 1 month, every 4 months during treatment period, and at the end of treatment (up to 5 years).
  The Brief Pain Inventory (BPI) questionnaire rapidly assesses the severity of pain and its impact on functioning. This self-report questionnaire includes:
  * A body schema
  * The maximum pain, lowest pain, usual pain within the last 15 days (Numeric rating scales (NRS) 0 to 10)
  * Description of current analgesic treatment,
  * An assessment of relief by a percentage scale (0-100%), Assessment of the impact of pain on: mood, relationships with others, walking, sleep, work, happiness the joy - of living, recreation, activities in general (digital scales, rating from 0 [normal] to 10 [no activity]).

CONTACTS AND LOCATIONS:
Overall Officials: Ronan FLIPPOT, MD, Principal Investigator — Gustave Roussy (Villejuif, France); David PASQUIER, MD, Principal Investigator — Centre Oscar Lambret, Lille University (Lille, France)
Locations (4):
- France (4):
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Centre Azuréen de Cancérologie, Mougins
  - CHU de Saint-Etienne, Saint-Etienne
  - Gustave Roussy Cancer Campus, Villejuif

IPD SHARING:
Plan to Share IPD: No